CLINICAL TRIAL: NCT01646580
Title: Study for the Assessment of Safety and Efficacy of Ciclopirox Olamine Cream in 3 Months to 10 Years Old Children With Dermatomycoses
Brief Title: Safety Study of Ciclopirox Olamine Cream for Dermatomycoses in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment rate. with the final sample primary endpoint could be assessed.
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CPO_08_01; 2008-003560-19 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Dermatomycoses
Keywords: dermatomycoses, tinea, candidiasis, children
MeSH Terms: conditions — Dermatomycoses; Tinea; Candidiasis | interventions — Ciclopirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ciclopirox (Experimental)
  Interventions: Drug: ciclopirox

INTERVENTIONS:
Drug: ciclopirox — Doses of 1.0% cream. Topical cream application. Twice daily for 28 days. Duration of treatment: 28 days with four weeks follow-up.
  Other Names: Ciclochem

SUMMARY:
Ciclopirox olamine (Ciclochem®) is a pyridone broad spectrum antifungal drug which has shown activity on dermatophytes, yeasts, moulds, actinomycetes and some bacteria. Its mechanism of action is based on a fungicidal activity by inhibiting the cellular captation of essential substances needed for the metabolism and growth of the fungi. On the other hand, this drug binds irreversibly with cell structures as mitochondria, ribosomes, microsomes and cell wall. After dermal application, Ciclopirox olamine undergoes skin penetration, being only absorbed a 1,5% of the applied dose. Clinical efficacy has been studied in patients above 10 years with superficial dermatomycoses (dermatophytoses, candidiasis and pityriasis versicolor) and the percentage of clinical healing ranged from 77% to 91% after 2-4 weeks of twice a day topical application. In all the studies, the safety profile has been very good, showing only a very low rate of adverse events of mild to moderate intensity. There are very few previous available data on the application of this compound in children under 10 years of age. A single study had been performed with a solution formulation in patients from 6 to 29 months with diaper candidiasis, showing good efficacy and tolerability in these patients. The present study aims to show the safety and tolerability of ciclopirox olamine in a cream formulation in patients from 3 months to 10 years with dermatomycoses.

DETAILED DESCRIPTION:
A multicenter, open, prospective, Phase IV study of Ciclopirox olamine on patients from 3 months to 10 years with all kinds of dermatomycoses. All body areas were treatable except scalp and nails (no tinea on the scalp nor onychomycoses) . Cream applied BID between 6.00 and 10.00am and 7.00 and 10.00pm daily for 4 weeks.Control visit after 4 more weeks without treatment was performed in order to evaluate the relapse rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 3 months to 10 years of age.
* Patients diagnosed of dermatomycoses produced by yeasts or dermatophytes by KOH technique at the inclusion moment, which has to be confirmed by culture.
* Obtention of the informed consent of the parents or legal representatives of the patients

Exclusion Criteria:

* Previous treatment with oral or topical antifungal drugs.
* Hypersensitivity to ciclopirox olamine or some of the cream excipients.
* Use of topical or oral steroids concomitantly.
* Patients with mycoses on the scalp or nails.

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To evaluate skin lesion condition as a measure of safety and tolerability of ciclopirox olamine treated dermatomycoses patients from 3 months to 10 years. | 28 days

SECONDARY OUTCOMES:
Explore clinical efficacy of topically applied ciclopirox olamine cream in patients with dermatomycoses. | 0, 7, 14, 21 and 28 days
Explore mycological efficacy of topically applied ciclopirox olamine cream in patients with dermatomycoses | 0, 7, 14, and 28 days
Explore relapse rate | day 56

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Moreno, Prof, PhD, Principal Investigator — Hospital Reina Sofia, Cordoba, Spain